CLINICAL TRIAL: NCT06139471
Title: Exploring the Efficacy of a Virtual Reality-Enhanced Gagne's Instructional Model in Promoting Nursing Students' Aging Rejection and Willingness Towards Gerontological Care
Brief Title: Efficacy of a Virtual Reality-Enhanced Gagne's Instructional Model
Acronym: VR-gagne
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 13-6-2021
Record Dates: First submitted 2023-11-02; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Acceptance Processes; Rejection, Psychology
Keywords: geriatric rejection; willingness towards Gerontological Care
MeSH Terms: conditions — Behavior; Rejection, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (VR-enhanced Gagne's Instructional Model) (Experimental): receive VR-enhanced Gagne's Instructional Model
  Interventions: Behavioral: Virtual Reality-Enhanced Gagne's Instructional Model
- STUDY group (No Intervention): doesn't VR-enhanced Gagne's Instructional Model

INTERVENTIONS:
Behavioral: Virtual Reality-Enhanced Gagne's Instructional Model — Virtual Reality-Enhanced Gagne's Instructional Model
  Arms: study group (VR-enhanced Gagne's Instructional Model)

SUMMARY:
Gagne's conditions of instructional learning theory, it presumed that several learning levels was exist that require different instruction types, and external and internal environments, commonly referred to as "conditions of learning".

DETAILED DESCRIPTION:
According to Robert Gagne's conditions of instructional learning theory, it presumed that several learning levels was exist that require different instruction types, and external and internal environments, commonly referred to as "conditions of learning", for every learning type. These internal conditions related to the learner's preexisting knowledge and external ones related to the instructions and teaching strategies provided by the instructor. The theory emphasizes the importance of both internal and external factors in creating a conducive learning environment that fosters effective learning outcomes According to this theorist, there are five primary knowledge categories, including verbal information, cognitive strategies, attitudes, and motor and intellectual skills.

ELIGIBILITY:
Inclusion Criteria:

1. Agreement to participate in this study.
2. Have a Microsoft team's account and able to use it.
3. No previous participation in any gerontological educational course either compulsory or elective.

exclusion Criteria: previous participation in any gerontological educational course either compulsory or elective.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Willingness to Work with Elderly People Scale (WEPS) | three months
  Nursing students who exposed to the VR-enhanced Gagne's Instructional Model will exhibit higher score in Willingness to Work with Elderly People Scale (WEPS) than who don't exposed to such therapy.

SECONDARY OUTCOMES:
The Fraboni Scale of Ageism (FSA) | 3 months
  Nursing students who exposed to the VR-enhanced Gagne's Instructional Model will exhibit lower score in The Fraboni Scale of Ageism (FSA) than who don't exposed to such therapy.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed H atta, Principal Investigator — Faculty of nursing, Alexandria university, Egypt
Locations (2):
- Egypt (2):
  - Mohamed Husien, Alexandria, Please Select A Country
  - Faculty of Nursing, Alexandria

IPD SHARING:
Plan to Share IPD: No